CLINICAL TRIAL: NCT04319666
Title: Intravascular Balloon Lithotripsy in Left Main Stem Percutaneous Coronary Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St George's, University of London (Other)
Collaborators: St George's University Hospitals NHS Foundation Trust (Other); Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019.0329
Record Dates: First submitted 2020-02-27; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Calcification; Left Main Coronary Artery Disease
Keywords: Coronary artery disease; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCI to left main with IVL (Experimental)
  Interventions: Device: Left main stenting with intravascular lithotripsy

INTERVENTIONS:
Device: Left main stenting with intravascular lithotripsy — Intravascular lithotripsy (IVL) will be used to modify coronary artery calcification prior to stent implantation in left main coronary disease. Intravascular ultrasound (IVUS) will be used pre and post IVL and post stenting.

SUMMARY:
The IVL Left Main study is a prospective non-randomised pilot study to investigate the mechanical and procedural outcomes and safety of distal left main stenting with coronary lithotripsy in addition to standard techniques in patients with calcific left main disease and a clinical indication for revascularisation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years old.
* Unprotected distal LM (or equivalent) disease defined as:

  1. >70% diameter stenosis (DS) on angiography in the distal LM; or
  2. ≥50% DS in the distal LM with a) non-invasive evidence of ischaemia referable to a hemodynamically significant left main lesion, and/or b) FFR ≤0.80; or
  3. >70% diameter stenosis in either the ostial left anterior descending (LAD) or ostial left circumflex (LCX) that is within 10 mm of the ostium and requires stenting back into the LM (distal LM equivalent); or
  4. >50% diameter stenosis in either the ostial left anterior descending (LAD) or ostial left circumflex (LCX) that is within 10 mm of the ostium and requires stenting back into the LM (distal LM equivalent) with a) non-invasive evidence of ischaemia referable to its myocardial territory and/or b) FFR ≤0.80
* Clinical indication for revascularisation by PCI
* Viability of the treatment vessel as determined by echocardiography, cardiac MRI or other equivalent imaging modality.
* ≥ 270° arc of calcification within at least one stenotic segment demonstrated on intravascular imaging.
* Ability to pass a 0.014" guide wire across the lesion.
* Ability to provide informed consent and comply with all study procedures, including follow-up at 30 days.
* Lesions not related to the distal LM requiring PCI can be treated:

  1. at the time of the study procedure if completed prior to distal LM PCI and the procedure was successful and uncomplicated (defined as a final lesion angiographic diameter stenosis <30% and TIMI 3 flow (visually assessed) for all non-target lesions and vessels without perforation, cardiac arrest or need for defibrillation or cardioversion or hypotension/heart failure requiring mechanical or intravenous hemodynamic support or intubation. In situations where the distal LM lesion is critical, the LM can be ballooned or treated first so long as the study protocol is not deviated.
  2. as a staged procedure either within the same hospital admission or within 30 days. Any staged procedure must be declared at the index procedure otherwise it will be recorded as an event.

Exclusion Criteria:

* Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.
* Daughter vessel reference diameter < 2.5 mm.
* Use of rotational atherectomy, scoring or cutting balloon, or any investigational device.
* Evidence of aneurysm in target vessel within 10 mm of the target lesion.
* Prior PCI of the LM or PCI of the proximal LAD or proximal LCX within 10 mm of the ostium.
* Prior coronary artery by-pass graft (CABG) surgery.
* Chronic total occlusion (CTO) of the LM, proximal LAD or proximal LCX.
* Untreated pre-procedural haemoglobin < 8 g/dL.
* Renal failure with serum creatinine > 2.5 mg/dL and not on chronic dialysis.
* Uncontrolled diabetes defined as a HbA1c >10%.
* Coagulopathy manifested by platelet count < 50,000/ mL or International Normalized ratio (INR) > 1.7 (INR is only required in patients who have taken warfarin within 2 weeks of enrolment).
* Cardiogenic shock.
* Ongoing ST elevation myocardial infarction (STEMI).
* History of stroke or transient ischemic attack (TIA) within 3 months.
* NYHA class IV heart failure or LVEF < 20%.
* Active peptic ulcer or upper gastrointestinal (GI) bleeding within 6 months.
* Patients with a life expectancy of less than 1 year.
* Visible thrombus (by angiography) at target lesion site.
* Patient has active systemic infection on the day of the index procedure with either fever or requiring intravenous antibiotics.
* Patient has vascular connective tissue disease (e.g. Marfan's syndrome).
* Patient has a hypercoagulable disorder.
* Patient has allergy to imaging contrast media for which they cannot be pre-medicated.
* Allergy to Aspirin.
* Allergy to Clopidogrel, Ticagrelor and Prasugrel.
* Allergy to any component of the drug eluting stent that is planned for use.
* Patient has any other severe comorbidity that is felt to preclude enrolment by the investigator.
* Subject is pregnant or nursing (a negative pregnancy test is required for women of child-bearing potential within 7 days prior to enrolment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary effectiveness endpoint 1 | Time of procedure
  Mean MSA (mm2) by segment for segments with obstructive disease and ≥ 270 degrees calcification.
Primary effectiveness endpoint 2 | Time of procedure
  Incidence of residual area stenosis <50% by segment for segments with obstructive disease and ≥ 270 degrees calcification.
Primary safety endpoint | 30 days
  Incidence of Major Adverse Cardiac Events (MACE) at 30 days MACE consists of cardiac death, myocardial infarction and target vessel revascularisation

SECONDARY OUTCOMES:
Minimum stent diameter (MSD) (mm) for segments with obstructive disease and ≥ 270 degrees calcification | Time of procedure
Stent symmetry ratio for segments with obstructive disease and ≥ 270 degrees calcification | Time of procedure
Stent expansion index (%) for segments with obstructive disease and ≥ 270 degrees calcification | Time of procedure
MSA (mm2) for all segments. | Time of procedure
MSD (mm) for all segments. | Time of procedure
Stent symmetry ratio for all segments. | Time of procedure
Stent expansion (%) for all segments. | Time of procedure
Device crossing success | Time of procedure
  ARC-2 criteria
Angiographic success | Time of procedure
  ARC-2 criteria
Procedural success | Time of procedure
  ARC-2 criteria
Serious angiographic complications | 24-48 hours
  ARC-2 criteria. Composite of loss of major vessel/side branch, embolisation, disruption of collateral flow, persistent slow-flow or no reflow, major dissection, new regional wall motion abnormality, imaging evidence of loss of viable myocardium.
MACE at 12 months | 12 months
Individual components of MACE at 30 days | 30 days
Individual components of MACE at 12 months | 12 months
Canadian Cardiovascular Society (CCS) angina status at 30 days | 30 days
Canadian Cardiovascular Society (CCS) angina status at 12 months | 12 months
Stroke at 30 days | 30 days
Stroke at 12 months | 12 months
Target lesion failure (TLF) at 30 days | 30 days
Target lesion failure (TLF) at 12 months | 12 months
Target vessel failure (TVF) at 30 days | 30 days
Target vessel failure (TVF) at 12 months | 12 months
All-cause mortality | 12 months
  Stratified by i) cardiac death ii) non-cardiac death
Peri-procedural myocardial infarction | 48 hours
  ARC-2 criteria
Spontaneous myocardial infarction | 12 months
  ARC-2 criteria
Ischaemic-driven revascularisation | 12 months
All revascularisation | 12 months
Angiographic and intracoronary imaging predictors of mechanical and procedural outcomes | 12 months
Correlation between CK-MB and/or troponin levels post-PCI and outcomes at 30-days and 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James Spratt, Principal Investigator — St George's University Hospitals NHS Foundation Trust
Locations (6):
- United Kingdom (6):
  - Belfast Health & Social Care Trust, Belfast, Northern Ireland
  - Golden Jubilee Hospital, Clydebank, Scotland
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - King's College Hospital NHS Foundation Trust, London
  - Royal Brompton & Harefield NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No